CLINICAL TRIAL: NCT05930951
Title: A Phase Ib Study of OBT076 or OBT076 Followed by Balstilimab in Patients With Recurrent or Metastatic (R/M) Adenoid Cystic Carcinoma (AdCC) of the Head and Neck (H&N)
Brief Title: Study of OBT076 Associated or Not in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma of the Head and Neck
Acronym: AdCC_2023-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: toxicity
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503270-20-00
Record Dates: First submitted 2023-06-23; First posted 2023-07-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Adenoid Cystic Carcinoma of the Head and Neck
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBT076 only (Active Comparator): OBT076, administration at 3mg/kg, (IV ≥ 3h infusion) on Day 1 every 21 days (3-week cycle) until disease progression, unacceptable toxicity, intercurrent conditions that preclude continuation of treatment or patient refusal whichever comes first.
  Interventions: Drug: OBT076
- OBT076 -Balstilimab (Experimental): 3 cycles of OBT076, administration at 3mg/kg, IV (≥ 3h infusion) on Day 1 every 21 days (3-week cycle) followed by Balstilimab, administration at 450mg, IV, on Day 1 every 21 days (3-week cycle) until disease progression, unacceptable toxicity, intercurrent conditions that preclude continuation of treatment or patient refusal whichever comes first.
  Interventions: Drug: OBT076; Drug: Balstilimab

INTERVENTIONS:
Drug: OBT076 — OBT076 is an ADC constituted by a fully human immunoglobulin 1 (IgG1) antibody directed against the CD205/Ly75 antigen (MBH1309), inducing potent cytotoxic and anti-tumor activity
Drug: Balstilimab — Balstilimab is a human monoclonal antibody that targets programmed cell death protein 1 (PD-1).
  Arms: OBT076 -Balstilimab

SUMMARY:
Adenoid cystic carcinoma (AdCC) is a rare salivary gland malignant tumor that accounts for approximately 1-3% of all head and neck cancers. AdCC is often charaterised by a long natural history with a propensity for indolent but relentless growth and dissemination. Local recurrences and late distant metastases are common findings in about 35% of the patients and associated with a poor prognosis1. AdCC is among the most lethal salivary gland tumors2 with no proven therapy for metastatic disease. Little is known about endogenous immune response directed against AdCC. However, in a relatively large series of 28 AdCC tumor, the immune profiling has shown in most tumors high and frequent programmed death ligand 2 (PD-L2) expression and PD-L1 was generally not expressed on tumor and infiltrating cells3.

The Antibody Drug Conjugates (ADCs) are emerging as a novel therapeutic option in cancer treatment that looks promising for solid tumors. An experimental CD205/Ly75-directed ADC, OBT076 induce potent cytotoxic and antitumor activity. Recently, the combination of immunohistochemistry (IHC) and tissue micro array (TMA) was performed in a series of 46 AdCC, showing a unique profile with both frequent and high expression of CD205/Ly75, much higher than for other solid tumors. In a phase I study, OBT076 demonstrated promising results for 3 patients with 2 partial responses and 1 complete response for a gastric cancer4. In this last patient, analysis showed an increase in PD1+, CD4+ and CD8+ cells suggesting that OBT076 activates the patient's immune response against the tumor, especially PD-1 targeted therapies4.

Based on this rational and on the high level of expression of CD205/Ly75 in AdCC, the hypothesis tested in this study is that OBT076 could be a potential effective treatment for R/M AdCC, which is an orphan lethal disease. The efficacy of OBT076 will be tested either alone or followed by an anti PD-1 inhibitor (Balstilimab) with the hypothesis that OBT076 will induce immune infiltrate that could restore sentivity to PD-1 targeting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female ≥ 18 years
2. ECOG PS 0-1
3. Histologically confirmed Adenoid Cystic Carcinoma (AdCC) of the Head and Neck or trachea
4. Histologically and/or radiologicaly documented recurrent or metastatic AdCC not amenable to surgery and/or radiotherapy
5. Patients with confirmed disease progression at study entry. The screening radiological evaluation (CT/MRI of H&N, chest, pelvis and brain if known or suspected cerebral involvement) should demonstrate disease progression according to RECIST 1.1 when compared to a prior disease assessment done within 6 months period prior to screening
6. Measurable disease by CT scan or MRI according to RECIST 1.1 criteria
7. Adequate haematologic, renal and hepatic function as indicated by (using CTCAE v5.0):

   * Absolute neutrophil count ≥ 2.0 × 109/L
   * Platelets ≥ 100 × 109/L
   * Hemoglobin ≥ 9.0 g/dL (blood transfusions during Screening are not permitted)
   * White blood cells ≥ 2 000/mm3
   * AST and ALT ≤ 2.5 × ULN in the absence of liver metastases or < 5 × ULN in the presence of liver metastases
   * Serum creatinine < 1.5 × ULN
   * Total bilirubin ≤ 1.5 × ULN (except Gilbert Syndrome < 3.0 mg/dL)
   * Potassium within normal range according to local lab, or correctable with supplements
8. The Investigator confirms that the participant agrees to use appropriate contraception and barriers methods, if applicable. The contraception, barrier, and pregnancy testing requirements are below:

   • A female participant: i. Is not a WOCBP, no need serum pregnancy test or contraceptive method ii. If WOCBP, she must agree to use a highly effective contraceptive method (i.e., with a failure rate of < 1% per year), preferably with low user dependency (as described in section 3.3), from ICF signature (ICF of the study not ICF of prescreening) to at least 4 months after the last dose of study drug. WOCBP must not agree to donate eggs (ova, oocytes) for reproduction during this period.

   • A male participant must agree to the following from ICF signature (ICF of the study not ICF of pre-screening) to at least 4 months after the last dose of study drug: i. To Refrain from donating fresh unwashed semen. If not done previously, cryopreservation of sperm prior to receiving study treatments is advised to male patients with a desire to have children. ii. Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use condom and spermicide. Because male condom and spermicide is not a highly effective contraception method, it is required that female partners of a male study participant use a highly effective contraceptive method (with a failure rate of < 1% per year).

   iii. If participants are sexually active, they must agree to use a highly effective contraceptive method (i.e., with a failure rate of < 1% per year), preferably with low user dependency
9. Patients with social insurance coverage
10. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the inform consent form and this protocol

Exclusion Criteria:

1. Pretreatment with a programmed cell death protein (PD-1), PD-L1 or cytotoxic T- lymphocyte antigen 4 (CTLA-4) therapy or any other immuno-checkpoint inhibitors.
2. Prior chemotherapy within 28 days before study drug administration.
3. Prior systemic anticancer therapy (regardless if approved or investigational therapy) within 5 halflives of study drug administration
4. Major surgery within 14 days before study drug administration
5. Patients have not recovered from the toxicities (CTCAE v5.0 grade > 1) of prior anticancer therapy
6. Prior curative radiotherapy ≤ 4 weeks or palliative radiotherapy ≤ 2 weeks before study drug administration, and/or from whom ≥ 30% of the bone marrow was irradiated
7. Patients with brain metastasis, except if treated with curative stereotactic radiotherapy
8. History of another malignancy within the last 2 years prior to randomization, with the exception of completely resected non-melanoma cell skin cancer outside the head and neck area or completely resected stage I breast cancer, gleason 6 localised prostate cancer, or completely resected in-situ non-muscular invasive bladder, cervix and/or uterine carcinomas.
9. Documented or suspected hypersensitivity or other contraindication to study drug or any excipients used in the manufacture of OBT076 or Balstilimab
10. Active or chronic corneal disorder or Sjogren's syndrome
11. Known history of infection with human immunodeficiency virus (HIV). If unknown history of HIV, an HIV screening test is to be performed and participants with positive serology for HIV-1/2 must be excluded.
12. Known chronically active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
13. Known active Covid 19 infection.
14. Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 28 days prior to study drug administration. The use of the inactivated seasonal influenza vaccine (Fluzone®) and covid vaccine is allowed.
15. Active or prior history of disease/medical condition listed below:

    * Known or underlying medical condition that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events
    * Subject has a past medical history of or ongoing clinically relevant interstitial lung disease, drug-induced pneumonitis or severe / very severe Chronic Obstructive Pulmonary Disease (COPD).
    * Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses (≤10 mg daily prednisone equivalent), are permitted in the absence of active autoimmune disease
    * Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years of the start of study treatment (i.e. with use of disease modifying agents or immunosuppressive drugs)
    * Ongoing uncontrolled infection requiring intravenous antibiotics, or requiring/ongoing oral antibiotics as continuation of a prior IV antibiotic course, antivirals or antifungals within 7 days prior to randomization Note: patients with localized fungal infection of skin or nails are eligible
16. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

    * Significant cardiac arrhythmia
    * Unstable angina or angina requiring surgical or medical intervention within 6 months prior to randomization
    * New York Heart Association Class > 2 congestive heart failure.
    * QTc using Fridericia's formula (QTcF) interval > 470 ms
17. Prior organ transplantation, including allogeneic stem cell transplantation
18. Pregnant or breastfeeding women
19. History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of drug administration.
20. Patient under guardianship, curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 1 year"
  ORR based on the best tumor response evaluated by investigator assessment using RECIST 1.1 criteria will be the primary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-André (Chu de Bordeaux), Bordeaux, France